CLINICAL TRIAL: NCT02334553
Title: Phase IIa, Placebo-controlled, Randomized, Double-blind, Crossover Single Dose Study to Evaluate the Safety, Tolerability and Efficacy of S-1226 (8%) Administered by Nebulization in Subjects With Mild Atopic Asthma.
Brief Title: Single Dose Study to Evaluate the Safety, and Efficacy of S-1226 (8%) in Subjects With Mild Atopic Asthma
Acronym: S-1226(8%)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SolAeroMed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SAMi-02-1-02
Record Dates: First submitted 2014-11-12; First posted 2015-01-08 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Asthma
Keywords: COPD; Chronic bronchitis; Cystic fibrosis; Bronchoconstriction; Perfluorocarbons; Carbon dioxide
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- S1226 (8%) (Active Comparator): The drug S1226(8%), consists of Perflubron and 8% CO2 in a medical gas mixture. The dosage is 3ml delivered as an aerosol/vapour/gas mixture with a Circulaire nebulizer.
  Interventions: Drug: S1226(8%)
- Placebo (Placebo Comparator): The comparator is normal saline delivered as an aerosol with compressed medical air with a Circulaire nebulizer.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S1226(8%) — The drug S1226(8%), consists of Perflubron (PFOB) and 8% CO2 delivered as an aerosol/vapour/gas mixture with a Circulaire nebulizer. The drug is administered as a single dose during the early phase asthmatic response for 2 minutes.
  Other Names: PFOB nebulized with 8% CO2 in medical gas mixture
  Arms: S1226 (8%)
Drug: Placebo — Normal saline nebulized with compressed medical air for 2 minutes during the early phase asthmatic response
  Other Names: normal saline nebulized with compressed medical air
  Arms: Placebo

SUMMARY:
Evaluate the safety and tolerability of a single dose of S-1226 (8%) in subjects with mild atopic asthma.

DETAILED DESCRIPTION:
Phase IIa, placebo-controlled, randomized, double-blind, crossover single dose study to evaluate the safety, tolerability and efficacy of S-1226 (8%) administered by nebulization in subjects with mild atopic asthma

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18-40 years of age.
2. BMI of 18-40 kg/m2
3. Subject is not currently on topical or systemic corticosteroids and has not taken any oral/injectable corticosteroid within 60 days prior to study drug administration and has not used any inhaled/nasal corticosteroid within 30 days prior to study drug administration.
4. Female subjects must not be pregnant or lactating and must be practicing an acceptable method of birth control, or be surgically sterile or postmenopausal.
5. Subjects must have had asthma for at least 3 months.
6. Subject is a non-smoker or has not smoked for > 1year and has < 10 pack-year history.
7. Subject has a methacholine PC20 of less than 16mg/mL.
8. Subject has normal laboratory values (normal values as clinically judged by the Investigator) for clinical chemistry, hematology, and urinalysis.
9. Subject is in general good health based on medical history and clinically acceptable results for the following assessments: physical examination, vital signs, and 12-lead ECG, as assessed by study physicians.
10. Subject is able to communicate effectively with study personnel and is reliable, willing and cooperative in terms of compliance with protocol.

Exclusion Criteria:

Subjects to whom any of the following applies will be excluded from the study:

1. Any clinically significant abnormality or abnormal laboratory test results found during medical screening or positive test for hepatitis B, hepatitis C, or HIV found during medical screening.
2. Subjects who require inhaled β2-agonist medication more frequently than 4 times a week (other than prophylactically prior to exercise) during the 4 week period before screening.
3. Subjects who are currently treated with any asthma medication other than inhaled β2-agonist.
4. Subjects with frequent emergency room visits for asthma, with prior ICU admission or those with prior intubation.
5. Presence or history of neurologic, endocrine, hepatic, gastrointestinal or kidney disease or therapy that would jeopardize the subject's well-being by participating in the study.
6. Cardiovascular disease that, in the opinion of the Investigator, is not stable or could put the subject at increased risk by participating in the study.
7. Any reason which, in the opinion of the Investigator (or delegate), would prevent the subject from participating in the study.
8. Clinically significant electrocardiogram (ECG) abnormalities or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
9. Subject has a history of physician diagnosed panic disorder or other anxiety disorders.
10. Subject is currently receiving treatment, or has received treatment in the previous 14 days, with monoamine oxidase (MAO) inhibitors.
11. Subjects dosed with an investigational drug within 30 days prior to the Screening Visit.
12. Subjects dosed with biologic therapy within the previous 4 months or 5 half-lives from baseline methacholine testing.
13. Subject has current (or within the last six months) evidence of alcohol abuse (regularly drinks more than 4 units of alcohol per day; 1 unit = ½ pint of beer, 1 glass of wine, or 1 ounce of spirit)
14. Positive urine drug screen or urine cotinine test at screening.
15. Breast-feeding subject.
16. Positive pregnancy test at screening.
17. Subject, who in the opinion of the Investigator, is mentally or emotionally unsuitable to participate, or unable/unwilling to comply with the study assessments.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-02-06 (Actual); Primary Completion 2015-11-25 (Actual); Study Completion 2015-11-25 (Actual)

PRIMARY OUTCOMES:
The number of treatment emergent adverse events (AEs). | 120 minutes
  Subjects will be closely monitored throughout the 2-minute drug and placebo administration periods and for 120 minutes following treatment. Treatment may be stopped at any time at the request of the subject and/or the qualified investigator or delegate.
  Safety and tolerability to S-1226 (8%) will be evaluated through the assessment of adverse events, vital signs, pulse oximetry, biochemistry and hematology testing, urinalysis, 12-lead ECG, physical examination, and pulmonary function (spirometry). These data will be recorded and descriptive statistics and change from baseline for safety parameters will be reported.

SECONDARY OUTCOMES:
Evaluate the efficacy of S-1226 (8%) in comparison to placebo. (evaluated using area under the curve (AUC) of the early asthmatic response (defined as a 20% fall from baseline FEV1 following allergen inhalation) | 30minutes
  Efficacy will be evaluated using area under the curve (AUC) of the early asthmatic response (defined as a 20% fall from baseline FEV1 following allergen inhalation), responder status which is achieving ≥ 25% reversal over placebo of the decrease in FEV1 from allergen challenge within 30 minutes after study treatment, maximum percent reversal of allergen-induced decrease in FEV1 in the first 30 minutes following study treatment administration, and the duration of the ≥ 25% reversal produced by study drug, defined as the interval after S-1226 (8%) administration during which the FEV1 is maintained at ≥ 25% above placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Leigh, MD, PhD, Principal Investigator — Professor and Head, Respiratory Clinical Trials Centre; Veronica Swystun, PhD, Study Director — Respiratory Clinical Trials Centre, University of Calgary
Locations (1):
- Respiratory Clinical Trials Centre, University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Background] El Mays TY, Choudhury P, Leigh R, Koumoundouros E, Van der Velden J, Shrestha G, Pieron CA, Dennis JH, Green FH, Snibson KJ. Nebulized perflubron and carbon dioxide rapidly dilate constricted airways in an ovine model of allergic asthma. Respir Res. 2014 Sep 16;15(1):98. doi: 10.1186/s12931-014-0098-x. PMID 25355286
- [Derived] Swystun V, Green FHY, Dennis JH, Rampakakis E, Lalli G, Fadayomi M, Chiu A, Shrestha G, El Shahat SG, Nelson DE, El Mays TY, Pieron CA, Leigh R. A phase IIa proof-of-concept, placebo-controlled, randomized, double-blind, crossover, single-dose clinical trial of a new class of bronchodilator for acute asthma. Trials. 2018 Jun 18;19(1):321. doi: 10.1186/s13063-018-2720-6. PMID 29914544
- See also: Pre clinical sheep model for S-1226 — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4172894/